CLINICAL TRIAL: NCT04270253
Title: End-range Mobilization Effecting Pain and Physical Function in the Management of Knee Osteoarthritis
Brief Title: End-range Mobilization on Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pecs (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PozsgaiMMaitlandKnee
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Osteo Arthritis Knee
Keywords: Musculoskeletal Manipulations; Osteoarthritis, Knee; Conservative Treatment
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Conservative Treatment; Musculoskeletal Manipulations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- End-range mobilization (Experimental): End-range mobilization applied 6 times for 2*2 min in end-range of flexion and extension end-range of the tibiofemoral and patellofemoral joint beside the same conservative therapy, as used for the Control
  Interventions: Procedure: Conservative therapy; Procedure: Manual therapy
- Control (Active Comparator): Conservative therapy including aquatic exercises (5-times), land-based exercises (3-times), balneotherapy (5-times) and TENS therapy (3-times)
  Interventions: Procedure: Conservative therapy

INTERVENTIONS:
Procedure: Conservative therapy — Conservative therapy including aquatic exercises, land-based exercises, balneotherapy, TENS therapy
Procedure: Manual therapy — End-range mobilization
  Arms: End-range mobilization

SUMMARY:
Different manual therapy techniques and conservative therapy have been used separately for alleviation of pain and improvement of physical function in patients with knee osteoarthritis (KOA). However, no study has reported the effect of combination of these treatment modalities in the management of KOA. The aim of this study was to investigate the effect of end-range mobilization added to conservative therapy versus conservative therapy alone on decrease of pain and improvement of functional status in KOA.

DETAILED DESCRIPTION:
Knee osteoarthritis (KOA) is a musculoskeletal condition affecting older people. It is characterized by pain and loss of physical function, which has a negative impact on patients' quality of life. The different international guidelines recommend several non-invasive treatment modalities for the management of KOA. Conservative therapy including land-based exercises, aquatic exercises, Transcutaneous Electro Neuro Stimulation (TENS) therapy and balneotherapy has been reported positively in the management of patients with KOA (1, 2). Manual therapy is also a preferred treatment modality with the aim of alleviation of pain, improvement of joint mobility and therefore the physical condition (1, 2). Out of manual therapy techniques, end-range mobilization is a well applied treatment technique in the management of different musculoskeletal conditions (3). Till date, the effect of end-range mobilization has not been investigated so far in knee OA.

Therefore, the aim of this study was to investigate the effect of end-range mobilization added to conservative therapy versus conservative therapy alone on decrease of pain and improvement of functional status in KOA.

ELIGIBILITY:
Inclusion Criteria:

* KOA according to the American College of Rheumatology
* categorization as End Of Range Problem based on Maitland's classification.
* at least half year existing and at least 3 pain scores measured with Visual Analogue Scale (VAS) during weight-bearing activities
* bilateral, moderate-to-severe symptomatic tibiofemoral knee OA with radiographic evidence
* at least 90 degree passive knee flexion range
* sufficient mental status

Exclusion Criteria:

* acute inflammation of the knee
* intraarticular injections within the last 3 months
* total knee replacement in the opposite side
* class II. obesity (body mass index, BMI>35kg/m2)
* severe degenerative lumbar spine disease (e.g. spondylolisthesis)
* systemic inflammatory arthritic or neurological condition
* physiotherapy and other balneotherapy attendance within 6 months
* contraindication for conservative and manual therapy
* unstable heart condition
* complex regional pain syndrome

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-05-12 (Actual)

PRIMARY OUTCOMES:
general pain intensity | at the end of the 3-week rehabilitation
  measuring of general pain intensity with Visual Analogue Scale

SECONDARY OUTCOMES:
pain intensity during getting up from a chair | at the end of the 3-week rehabilitation
  measuring of pain intensity during getting up from a chair with Visual Analogue Scale
pain intensity during getting in car | at the end of the 3-week rehabilitation
  measuring of pain intensity during getting in car with Visual Analogue Scale
pain intensity during turning while walking | at the end of the 3-week rehabilitation
  measuring of pain intensity during turning while walking with Visual Analogue Scale
pain intensity during stair descending | at the end of the 3-week rehabilitation
  measuring of pain intensity during stair descending with Visual Analogue Scale
Flexion and extension passive range of motion | at the end of the 3-week rehabilitation
  Flexion and extension passive range of motion of the tibiofemoral joint
Quadriceps and hamstring muscles peak muscle force | at the end of the 3-week rehabilitation
  Quadriceps and hamstring muscles peak muscle force of both knees
6-minute walk test | at the end of the 3-week rehabilitation
  6-minute walk test measuring functional capacity
Timed Up and Go test | at the end of the 3-week rehabilitation
  Timed Up and Go test measuring functional capacity

CONTACTS AND LOCATIONS:
Overall Officials: Miklós Pozsgai, Study Chair — Zsigmondy Vilmos Spa and Balneological Hospital of Harkány
Locations (1):
- Zsigmondy Vilmos Spa and Balneological Hospital of Harkány, Harkány, Please Select, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hochberg MC, Altman RD, April KT, Benkhalti M, Guyatt G, McGowan J, Towheed T, Welch V, Wells G, Tugwell P; American College of Rheumatology. American College of Rheumatology 2012 recommendations for the use of nonpharmacologic and pharmacologic therapies in osteoarthritis of the hand, hip, and knee. Arthritis Care Res (Hoboken). 2012 Apr;64(4):465-74. doi: 10.1002/acr.21596. PMID 22563589
- [Background] McAlindon TE, Bannuru RR, Sullivan MC, Arden NK, Berenbaum F, Bierma-Zeinstra SM, Hawker GA, Henrotin Y, Hunter DJ, Kawaguchi H, Kwoh K, Lohmander S, Rannou F, Roos EM, Underwood M. OARSI guidelines for the non-surgical management of knee osteoarthritis. Osteoarthritis Cartilage. 2014 Mar;22(3):363-88. doi: 10.1016/j.joca.2014.01.003. Epub 2014 Jan 24. PMID 24462672
- [Background] Maricar N, Shacklady C, McLoughlin L. Effect of Maitland mobilization and exercises for the treatment of shoulder adhesive capsulitis: a single-case design. Physiother Theory Pract. 2009 Apr;25(3):203-17. doi: 10.1080/09593980902776654. PMID 19384739